CLINICAL TRIAL: NCT06317649
Title: A Randomized Phase II Study of Venetoclax and HMA-Based Therapies for the Treatment of Older and Unfit Adults With Newly Diagnosed FLT3-Mutated Acute Myeloid Leukemia (AML): A MyeloMATCH Treatment Trial
Brief Title: Venetoclax and HMA Treatment of Older and Unfit Adults With FLT3 Mutated Acute Myeloid Leukemia (AML) (A MyeloMATCH Treatment Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01987; NCI-2024-01987 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MM1OA-EA02 (Other: ECOG-ACRIN Cancer Research Group); MM1OA-EA02 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-03-16; First posted 2024-03-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Specimen Handling; Biopsy; gilteritinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Regimen 1 (azacitidine, venetoclax) (Experimental): INDUCTION: Patients receive azacitidine IV or SC on days 1-7 of each cycle and venetoclax PO on days 1-28 of each cycle. Treatment repeats every 28 days for up to 2 cycles or until patient achieves remission, whichever comes first, in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients receive azacitidine IV or SC on days 1-7 and venetoclax PO on days 1-28 of each cycle. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Patients undergo bone marrow biopsy and aspiration as well as blood sample collection on the trial.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Venetoclax
- Regimen 2 (azacitidine, venetoclax, gilteritinib) (Experimental): INDUCTION: Patients receive azacitidine IV or SC on days 1-7 and venetoclax and gilteritinib PO on days 1-28 of each cycle. Treatment repeats every 28 days for up to 2 cycles or until patient achieves remission, whichever comes first, in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients receive azacitidine IV or SC on days 1-5, venetoclax PO on days 1-7 and gilteritinib PO on days 1-28 of each cycle. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Patients undergo bone marrow biopsy and aspiration as well as blood sample collection on the trial.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Gilteritinib; Drug: Venetoclax
- Regimen 3 (azacitidine, venetoclax, gilteritinib) (Experimental): INDUCTION: Patients receive azacitidine IV or SC on days 1-7 and venetoclax PO on days 1-28, and gilteritinib PO on days 8-21 of each cycle. Treatment repeats every 28 days for up to 2 cycles or until patient achieves remission, whichever comes first, in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients receive azacitidine IV or SC on days 1-5, venetoclax PO on days 1-14 and gilteritinib PO on days 8-21 of each cycle. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Patients undergo bone marrow biopsy and aspiration as well as blood sample collection on the trial.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Gilteritinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Gilteritinib — Given PO
  Other Names: ASP 2215; ASP-2215; ASP2215
  Arms: Regimen 2 (azacitidine, venetoclax, gilteritinib); Regimen 3 (azacitidine, venetoclax, gilteritinib)
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II MyeloMATCH treatment trial compares the usual treatment of azacitidine and venetoclax to the combination treatment of azacitidine, venetoclax and gilteritinib in treating older and unfit patients with acute myeloid leukemia and FLT3 mutations. Azacitidine is a drug that is absorbed into DNA and leads to the activation of cancer suppressor genes, which are genes that help control cell growth. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Gilteritinib is in a class of medications called kinase inhibitors. It works by blocking the action of a certain naturally occurring substance that may be needed to help cancer cells multiply. This study may help doctors find out if these different approaches are better than the usual approaches. To decide if they are better, the study doctors are looking to see if the study drugs lead to a higher percentage of patients achieving a deeper remission compared to the usual approach.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the achievement rate of measured residual disease negative (MRDneg) complete remission (CR) of either triplet regimen to azacitidine and venetoclax alone within 4 cycles of therapy.

SECONDARY OBJECTIVES:

I. To compare the achievement rate of MRDneg CR/complete remission with incomplete count recovery (CRi)/complete remission with partial hematologic recovery (CRh) of either triplet regimen to azacitidine and venetoclax alone within 4 cycles of therapy.

II. To determine the safety and tolerability of the combination of gilteritinib, azacitidine, and venetoclax, if both of the triplet regimens show superiority to the azacitidine plus venetoclax regimen.

III. To determine the optimal sequence and duration of gilteritinib, when added to azacitidine and venetoclax if both of the triplet regimens show superiority to the azacitidine plus venetoclax regimen.

IV. To estimate the rates of complete remission (CR), complete remission with incomplete count recovery (CRi), and complete remission with partial hematologic recovery (CRh), morphologic leukemia-free state (MLFS), event-free survival (EFS), and overall survival (OS) of the combination of gilteritinib, azacitidine, and venetoclax versus azacitidine and venetoclax alone.

EXPLORATORY OBJECTIVES:

I. To establish the degree reduction in FLT3- internal tandem duplication (ITD) mutation burden after 2 and 4 cycles of therapy using a highly sensitive next-generation sequencing (NGS) MRD assay and compare the median reduction in the investigational regimens among patients with CR/CRi/CRh to that of control regimen.

II. To determine if the degree of FLT3 ITD reduction is associated with the duration of remission.

III. To monitor which mutations are present at the time of relapse. IV. To monitor which co-mutations at presentation are associated with lack of response to these regimens.

V. To determine if the FLT3 AR /variant allele frequency (VAF) is associated with response to the regimens.

OUTLINE: Patients are randomized to 1 of 3 regimens.

REGIMEN 1:

INDUCTION: Patients receive azacitidine intravenously (IV) or subcutaneously (SC) on days 1-7 of each cycle and venetoclax orally (PO) on days 1-28 of each cycle. Treatment repeats every 28 days for up to 2 cycles or until patient achieves remission, whichever comes first, in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients receive azacitidine IV or SC on days 1-7 and venetoclax PO on days 1-28 of each cycle. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

REGIMEN 2:

INDUCTION: Patients receive azacitidine IV or SC on days 1-7 and venetoclax and gilteritinib PO on days 1-28 of each cycle. Treatment repeats every 28 days for up to 2 cycles or until patient achieves remission, whichever comes first, in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients receive azacitidine IV or SC on days 1-5, venetoclax PO on days 1-7 and gilteritinib PO on days 1-28 of each cycle. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

REGIMEN 3:

INDUCTION: Patients receive azacitidine IV or SC on days 1-7 and venetoclax PO on days 1-28, and gilteritinib PO on days 8-21 of each cycle. Treatment repeats every 28 days for up to 2 cycles or until patient achieves remission, whichever comes first, in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients receive azacitidine IV or SC on days 1-5, venetoclax PO on days 1-14 and gilteritinib PO on days 8-21 of each cycle. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

All patients undergo bone marrow biopsy and aspiration as well as blood sample collection on the trial.

After completion of study treatment, patients are followed up every 3 months if patient is < 2 years from first registration, and every 6 months if patient is 2-5 years from first registration. All patients, including those who discontinue protocol therapy early, are followed for response until progression, even if non-protocol therapy is initiated, and for survival for 10 years from the date of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 60 years of age or adults ˂ 60 who in the opinion of the treating physician are better served by azanucleoside-based therapy rather than intensive, cytarabine-based induction based on clinical status (i.e., performance status, age > 75 years), organ dysfunction, or disease biology
* Patient must have a morphologically confirmed diagnosis of AML according to the World Health Organization (WHO) 2016 classification excluding acute promyelocytic leukemia (APL) with PML-RARA, AML with RUNX1-RUNX1T1, or AML with CBFB-MYH11
* Patient must have no prior therapy for AML with the exception of hydroxyurea and all-trans retinoic acid (ATRA), or leukapheresis. Patients with cytarabine-based emergency therapy prior to the start of therapy on this trial are eligible
* Patient must have no prior therapy with hypomethylating agents or FLT3 inhibitors
* Patient must have the FLT3-ITD or D835 mutation based on MyeloMATCH Master Screening and Reassessment Protocol (MSRP)
* Patient must be assigned to this protocol by the myeloMATCH MSRP
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used.

  * All patients of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy.
  * A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient of childbearing potential and/or sexually active patients must not expect to conceive or father children by using an accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study. Contraception measures must continue for 30 days after the last dose of venetoclax for all patients and for 6 months after the last dose of gilteritinib for patients of childbearing potential and for 4 months after the last dose of gilteritinib for male patients with partners of childbearing potential. Patient must not breastfeed during treatment and for 2 months after treatment ends
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* Total bilirubin 2X ≤ institutional upper limit of normal (ULN) (unless thought to be elevated due to disease involvement or Gilbert's syndrome)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional ULN

  * Either measured or estimated by Cockcroft-Gault equation
* Creatinine clearance of ≥ 30 mL/min/1.73m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration/randomization are eligible for this trial
* Patients must not have a baseline corrected QT interval ≥ 480 msec using Fredericia correction (QTcF).

NOTE: Since older patients are at risk for prolonged QTc and many will require supportive care with agents that affect the QTc, an ECG is recommended if clinically indicated. If the QTc is prolonged, they should be treated on tier advancement process (TAP) instead of EA02

* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patient must not have the medical necessity for ongoing treatment with a strong CYP3A4 inducing drug
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients must not have an active or uncontrolled infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2029-05-15 (Estimated); Study Completion 2029-05-15 (Estimated)

PRIMARY OUTCOMES:
Rate of measured residual disease (MRD) negative complete remission (CR) | Up to 4 cycles of treatment
  Will be assessed by multiparameter flow cytometry at a level of ≤ 1 residual blast / 1,000 leukocytes (≤ 10^-3).

SECONDARY OUTCOMES:
Overall survival | Time between randomization and death from any cause, assessed up to 10 years
  Will be calculated using the Kaplan-Meier method.
Event-free survival | Time from randomization to failure to achieve complete remission (CR), CR with incomplete count recovery, and CR with partial hematologic recovery, or to relapse after CR/CRi/CRh or to death in remission, assessed up to 10 years
  Will be calculated using the Kaplan-Meier method.
Incidence of adverse events | Up to 10 years
  Will be determined using the Common Terminology Criteria for Adverse Events version 5 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica K Altman, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (213):
- United States (211):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Mills Health Center, San Mateo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Yale University, New Haven, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - MaineHealth Cancer Care and IV Therapy - Brunswick, Brunswick, Maine
  - Mid Coast Hospital, Brunswick, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - George E Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Puerto Rico (2):
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm